CLINICAL TRIAL: NCT00003917
Title: An Open Label, Multicenter, Randomized, Phase III Comparator Study of Oral Topotecan Versus Intravenous Topotecan for Second Line Therapy in Patients With Small Cell Lung Cancer Who Have Relapsed Greater Than or Equal to 90 Days After Completion of First Line Therapy
Brief Title: Topotecan in Treating Patients With Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Smith Kline Beecham (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: SKF1598; CWRU-SKF-1598; SB-104864-A/396; NCI-G99-1524
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if topotecan is more effective given by infusion or by mouth.

PURPOSE: Randomized phase III trial to compare the effectiveness of topotecan given by infusion with that of topotecan given by mouth in treating patients who have small cell lung cancer that has relapsed following previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the response rate, response duration, time to response, time to progression, and survival of patients with relapsed limited or extensive stage small cell lung cancer treated with oral vs intravenous topotecan. II. Compare the qualitative and quantitative toxicities of these treatment regimens in this patient population. III. Compare the quality of life in these patients.

OUTLINE: This is randomized, multicenter study. Patients are stratified according to gender, liver metastases (yes vs no), and duration of response to prior chemotherapy (6 months or less vs greater than 6 months). Patients are randomized to one of two treatment arms. Arm I: Patients receive topotecan IV over 30 minutes on days 1-5. Arm II: Patients receive topotecan orally on days 1-5. Treatment repeats every 3 weeks in the absence of unacceptable toxicity. Patients experiencing complete or partial response continue until progression or for at least 2 courses past maximal response. Patients with stable disease should receive at least 4 courses. Quality of life is assessed Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 300 patients (150 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed limited or extensive stage small cell lung cancer (SCLC) Disease recurring at least 90 days following completion of first line chemotherapy Partial or complete response to first line therapy Must have at least one bidimensionally measurable non CNS lesion May be within a prior radiation port if at least 6 weeks since prior radiotherapy and progressing Brain and/or leptomeningeal metastases allowed if asymptomatic and not requiring corticosteroids

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 2 months Hematopoietic: WBC at least 3,500/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL (after transfusion, if needed) Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT and SGPT no greater than 2 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present) Alkaline phosphatase no greater than 2 times ULN (no greater than 5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: No active uncontrolled infection No other malignancies within the past 5 years except curatively treated basal or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I low grade prostate cancer No other severe medical conditions that would preclude study or cause exposure to extreme risk or decreased life expectancy No uncontrolled emesis No active peptic ulcer, diabetes mellitus, chronic gastritis, significant ascites, or other gastrointestinal (GI) conditions (e.g., removal of a portion of the stomach or recent GI obstruction) that would alter absorption or GI motility No history of allergic reactions to compounds chemically related to topotecan Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception for 3 months prior to, during, and at least 4 weeks after the study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 months since prior immunotherapy No concurrent immunotherapy for SCLC Chemotherapy: See Disease Characteristics No prior topotecan Only one prior chemotherapy regimen allowed No other concurrent chemotherapy for SCLC Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics At least 24 hours since prior radiotherapy No concurrent radiotherapy for SCLC Surgery: At least 4 weeks since prior surgery Other: At least 30 days or five half lives since other prior investigational drugs No prior drugs (e.g., cisapride) that would alter absorption or GI motility No other concurrent investigational therapy for SCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 1999-03; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Levitan, MD, Study Chair — Case Comprehensive Cancer Center
Locations (53):
- United States (53):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Pacific Coast Hematology/Oncology Medical Group, Fountain Valley, California
  - Scripps Clinic, La Jolla, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Southwest Cancer Care, Poway, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Sidney Kimmel Cancer Center, San Diego, California
  - Oncology Clinic, P.C., Colorado Springs, Colorado
  - Shands Cancer Center, Gainesville, Florida
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Baptist Hospital- Pensacola, Pensacola, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Medical College of Georgia Hospital and Clinics, Augusta, Georgia
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Oncology and Hematology Associates, Inc., Indianapolis, Indiana
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Alton Ochsner Medical Foundation Hospital, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - St. Joseph Mercy Hospital, Pontiac, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Cooper Cancer Institute, Camden, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Cooper Hospital/University Medical Center, Voorhees Township, New Jersey
  - Santa Fe Hematology/Oncology, Santa Fe, New Mexico
  - Rochester General Hospital, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Salem Research, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Central Pennsylvania Hematology & Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Brown University Oncology Group, Providence, Rhode Island
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - Sarah Cannon-Minnie Pearl Cancer Center, Nashville, Tennessee
  - Texas Cancer Care, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Office of Michael E. Lee, Norfolk, Virginia
  - Hematology & Oncology Associates of Virginia, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Waukesha Memorial Hospital, Waukesha, Wisconsin

REFERENCES:
- [Result] Eckardt JR, von Pawel J, Pujol JL, Papai Z, Quoix E, Ardizzoni A, Poulin R, Preston AJ, Dane G, Ross G. Phase III study of oral compared with intravenous topotecan as second-line therapy in small-cell lung cancer. J Clin Oncol. 2007 May 20;25(15):2086-92. doi: 10.1200/JCO.2006.08.3998. PMID 17513814